CLINICAL TRIAL: NCT06581718
Title: Eye Gaze Technology for Endoscopic Inspection of the Gastrointestinal Tract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20SM6304
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cancer Gi
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Gaze (Experimental)
  Interventions: Device: Eye Gaze Control

INTERVENTIONS:
Device: Eye Gaze Control — Eye Gaze Control - UGI and LGI endoscopy

SUMMARY:
Robotic controlled endoscopy of GI tract.

DETAILED DESCRIPTION:
A robotised conventional endoscope will be used to examine the GI tract of 10 patients following successful benchtop trials.

ELIGIBILITY:
Inclusion Criteria:

* Routine UGI endoscopic indications

Exclusion Criteria:

* Varices
* <18
* GI haemorrhage
* PS > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Time of completion | 6 months
User Experience survey | 6 months
Patient Experience survey | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, Lonodon, United Kingdom

IPD SHARING:
Plan to Share IPD: No